CLINICAL TRIAL: NCT01163422
Title: Long-term Right Ventricular Resynchronization Therapy for Chronic Thromboembolic Pulmonary Hypertension
Brief Title: Right Ventricular Resynchronization Therapy
Acronym: RVRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Hanno L. Tan, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MEC 09/307
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2009-12

CONDITIONS: Right Ventricular Failure; Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Hypertension
Keywords: Right ventricular failure; Pacemaker; Cardiac resynchronization therapy; Pulmonary hypertension
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate RVRT (Active Comparator): RVRT switched on immediately after pacemaker implant
  Interventions: Device: Implantation of 3-chamber pacemaker
- Delayed RVRT (Placebo Comparator): RVRT switched on 4 weeks after pacemaker implant
  Interventions: Device: Implantation of 3-chamber pacemaker

INTERVENTIONS:
Device: Implantation of 3-chamber pacemaker — Implantation of pacemaker with leads in right atrium, right ventricle, and coronary sinus (left ventricle) with the aim of providing right ventricular resynchronization therapy (RVRT); this is accomplished by pacing the right ventricle ahead of the left ventricle, e.g., by setting (shortening) the A-V delay between right atrium and right ventricle to an optimal level.
  Other Names: Medtronic CRT pacemaker systems will be implanted

SUMMARY:
The purpose of this study is to determine whether cardiac resynchronization therapy with the use of an implanted electronic pacemaker reduces morbidity associated with chronic thromboembolic pulmonary hypertension

DETAILED DESCRIPTION:
Rationale: The clinical severity of right ventricular disease is largely determined by right-to-left ventricular dyssynchrony, i.e., delay of electrical activity between the right and left ventricles. Moreover, in patients with chronic thromboembolic pulmonary hypertension (CTEPH), we found that acute correction of this dyssynchrony by temporary pacing (prior to pulmonary endarterectomy, presently the therapy of choice for CTEPH) results in significant improvement in cardiac output. In this study, we aim to establish whether chronic pacing with the use of implanted pacemakers confers long-lasting improvements in cardiac output and functional class.

Objective: To study whether chronic pacing with implanted pacemakers confers long-lasting improvements in cardiac output and functional class in severely symptomatic CTEPH patients who are not eligible for pulmonary endarterectomy, or those in whom pulmonary endarterectomy has failed.

Study design: Chronic intervention study, double-blinded, randomized, cross-over.

Study population: Adult CTEPH patients who are not eligible for pulmonary endarterectomy, or those in whom pulmonary endarterectomy has failed.

Intervention (if applicable): chronic right ventricular resynchronization therapy (RVRT), i.e., chronic right atrial, right ventricular, and left ventricular pacing with the use of implanted pacemakers.

Main study parameters/endpoints: (Duration of) improvements (in l/min) in cardiac output as measured using Doppler echocardiography, and functional class as measured using 6-minute walking distance (6-MWD), right and left ventricular dimensions and ejection fractions (99mTechnetium scintigraphy), biomarkers for heart failure (serum NT-proBNP levels), and quality of life (SF-36) questionnaire.

Design: Randomized, double-blind, cross-over study with 2 arms of 10 patients each (arms 1 and 2). In arm 1, RVRT is switched on immediately after pacemaker implant, is switched of in week 5, and switched on at the start of week 6 until study end (32 weeks). In arm 2, RVRT is switched at the start of week 5 after pacemaker implant until study end (32 weeks). At various follow-up visits at weeks 1, 4, 5, 6, 8, 12, 16, the main study parameters/endpoints (see previous paragraph) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with chronic thromboembolic pulmonary hypertension (CTEPH) who are ineligible for pulmonary endarterectomy, and those in whom pulmonary endarterectomy has failed

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in right/left ventricular synchrony measured using tissue Doppler echocardiography | within 8 months after pacemaker implantation
Increase in cardiac output measured using Doppler echocardiography and scintigraphy | within 8 months after pacemaker implantation
Increase in functional capacity measured with six-minute walking distance | within 8 months after pacemaker implantation

SECONDARY OUTCOMES:
Increase in well-being assessed with questionnaire | within 8 months after pacemaker implantation

CONTACTS AND LOCATIONS:
Overall Officials: Hanno L Tan, MD,PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, University of Amsterdam, Amsterdam, Netherlands